CLINICAL TRIAL: NCT00003234
Title: A Phase II Study of Navelbine (Vinorelbine) In Children With Recurrent Or Refractory Malignancies
Brief Title: Vinorelbine in Treating Children With Recurrent or Refractory Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: A09705; COG-A09705 (Other: Children's Oncology Group); CCG-09705 (Other: Children's Cancer Group); CDR0000066106 (Other: Clinical Trials.gov)
Record Dates: First submitted 1999-11-01; First posted 2003-10-28 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Brain and Central Nervous System Tumors; Neuroblastoma; Sarcoma
Keywords: recurrent childhood rhabdomyosarcoma; recurrent neuroblastoma; recurrent childhood soft tissue sarcoma; recurrent childhood supratentorial primitive neuroectodermal tumor; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent childhood ependymoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Neuroblastoma; Sarcoma; Astrocytoma; Neuroectodermal Tumors, Primitive, Peripheral; Familial ependymoma | interventions — Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Stratum 1 - Soft Tissue Sarcoma (Experimental): See detailed description.
  Interventions: Drug: vinorelbine tartrate
- Stratum 2 - CNS Tumors (Experimental): See detailed description.
  Interventions: Drug: vinorelbine tartrate
- Stratum 3 - Neuroblastoma (Experimental): See detailed description.
  Interventions: Drug: vinorelbine tartrate

INTERVENTIONS:
Drug: vinorelbine tartrate
  Other Names: Navelbine®; 3',4'-didehydro-4'-deoxy-C'-norvincaleukoblastine [R-(R*,R*)-2,3,-dihydroxybutanedioate)

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of vinorelbine in treating children with recurrent or refractory cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate of children with recurrent or refractory malignancies treated with vinorelbine. II. Assess the toxic effects of this drug in these children.

OUTLINE: Patients receive vinorelbine IV over 6-10 minutes weekly on weeks 1-6. Treatment repeats every 8 weeks for a total of 10 courses in the absence of disease progression or unacceptable toxicity. Patients are followed every 4 months for 2 years, every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A maximum of 100 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed recurrent or refractory solid malignant tumors of childhood including: Soft tissue sarcoma Rhabdomyosarcoma Nonrhabdomyosarcoma Extraosseous Ewing's sarcoma CNS tumors Astrocytoma Primitive neuroectodermal tumor Atypical teratoid/rhabdoid tumors Ependymoma Recurrent neuroblastoma Measurable disease No more than 2 prior treatment regimens

PATIENT CHARACTERISTICS: Age: 21 and under at diagnosis Performance status: ECOG 0-2 Life expectancy: At least 2 months Hematopoietic: For patients with solid tumors (unless marrow involvement): Absolute neutrophil count (ANC) at least 1000/mm3 Platelet count at least 100,000/mm3 (transfusion independent) Hemoglobin at least 10 g/dL (RBC transfusions allowed) For patients post bone marrow transplantation: ANC at least 1,000/mm3 Platelet count at least 50,000/mm3 (transfusion independent) Hemoglobin at least 10 g/dL (RBC transfusions allowed) Hepatic: Total bilirubin no greater than 1.5 times normal SGOT/SGPT less than 2.5 times normal Renal: Creatinine no greater than 1.5 times normal OR Creatinine clearance or radioisotope glomerular filtration rate at least 70 mL/min Neurologic: Seizure disorder allowed if well controlled CNS toxicity no greater than grade 2

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 6 months since prior bone marrow transplantation No concurrent immunomodulating agents Chemotherapy: At least 2 weeks since prior chemotherapy (4 weeks for nitrosourea) and recovered No other concurrent chemotherapy Endocrine therapy: No concurrent corticosteroids except for increased intracranial pressure due to CNS tumors Radiotherapy: At least 6 months since prior radiotherapy to craniospinal axis, spine, and/or more than 50% of the bony pelvis Concurrent radiotherapy to localized painful lesions allowed if at least one measurable lesion is not in radiation field Surgery: Not specified Other: No concurrent participation in another CCG, POG, or COG therapeutic study

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 1998-05; Primary Completion 2006-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Disease progression

CONTACTS AND LOCATIONS:
Overall Officials: John F. Kuttesch, PhD, MD, Study Chair — M.D. Anderson Cancer Center
Locations (228):
- United States (200):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - University of South Alabama Medical Center, Mobile, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - University of California San Diego Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Jonathan Jaques Children's Cancer Center, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Children's Hospital of Oakland, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital at Stanford, Palo Alto, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Medical Center, Sacramento, California
  - Kaiser Permanente-Southern California Permanente Medical Group, San Diego, California
  - Children's Hospital and Health Center, San Diego, California
  - Kaiser Permanente Medical Group - San Francisco, San Francisco, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Childhood Hematology/Oncology Associates, Denver, Colorado
  - Children's Hospital of Denver, Denver, Colorado
  - Presbyterian-St Luke's Medical Center, Denver, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Alfred I. Dupont Institute, Wilmington, Delaware
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Shands Hospital and Clinics, University of Florida, Gainesville, Florida
  - Joe DiMaggio Children's Hospital at Memorial, Hollywood, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami-Jackson Memorial Hospital Medical Center, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Walt Disney Memorial Cancer Institute, Orlando, Florida
  - Nemours Children's Clinic-Orlando, Orlando, Florida
  - Sacred Heart Children's Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Tampa Children's Hospital, Tampa, Florida
  - St. Mary's Hospital, West Palm Beach, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Children's Healthcare of Atlanta - Scottish Rite, Atlanta, Georgia
  - Medical College of Georgia Comprehensive Cancer Center, Augusta, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Memorial Health University Medical Center, Inc., Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Mountain States Tumor Institute, Boise, Idaho
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Children's Memorial Hospital, Chicago, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Hope Children's Hospital, Oak Lawn, Illinois
  - Lutheran General Hospital, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - University Child Health Services Clinic, Rockford, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - St. Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Raymond Blank Memorial Hospital for Children, Des Moines, Iowa
  - John Stoddard Cancer Center, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - Wesley Medical Center, Wichita, Kansas
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Ochsner Clinic, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Boston Floating Hospital Infants and Children, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - St. John Hospital and Medical Center, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Spectrum Health and DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Duluth Clinic, Duluth, Minnesota
  - Children's Hospitals and Clinics - Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Children's Hospitals and Clinics of Minnesota, Saint Paul, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Children's Hospital of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - Atlantic Health System, Summit, New Jersey
  - University of New Mexico School of Medicine, Albuquerque, New Mexico
  - Cancer Center of Albany Medical Center, Albany, New York
  - Brooklyn Hospital Center, Brooklyn, New York
  - State University of New York Health Science Center at Brooklyn College of Medicine, Brooklyn, New York
  - Brookdale University Hospital and Medical Center, Brooklyn, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Columbia Presbyterian Hospital, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Saint Joseph's Health System, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Healthcare, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - Dakota Cancer Institute, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Children's Hospital of Columbus, Columbus, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Toledo Children's Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Forum Health-Tod Childrens Hospital, Youngstown, Ohio
  - Children's Hospital of Oklahoma, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center, Tulsa, Oklahoma
  - Doernbecher Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Center for Cancer Treatment and Research, Columbia, South Carolina
  - Children's Hospital of Greenville Hospital System, Greenville, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sioux Valley Hospital, Sioux Falls, South Dakota
  - James H. Quillen College of Medicine, Johnson City, Tennessee
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine, Amarillo, Texas
  - Children's Hospital of Austin, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - San Antonio Military Pediatric Cancer and Blood Disorders Center, Lackland Air Force Base, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - Methodist Health Care System, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Vermont Cancer Center, Burlington, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Massey Cancer Center, Richmond, Virginia
  - Carilion Roanoke Community Hospital, Roanoke, Virginia
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Cooperative of Puget Sound, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Mary Bridge Children's Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University - Charleston, Charleston, West Virginia
  - Cabell-Huntington Hospital, Inc, Huntington, West Virginia
  - West Virginia University Hospitals, Morgantown, West Virginia
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (5):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital, Brisbane, Queensland
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (16):
  - Alberta Children's Hospital, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Children's Health and Rehabilitation Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - Children's Hospital, Hamilton, Ontario
  - Children's Hospital of Western Ontario, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - McGill University Health Center - Montreal Children's Hospital, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Laval University Medical Center, Sainte-Foy, Quebec
  - Centre Hospitalier de L'Universite Laval, Sainte-Foy, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Academisch Ziekenhuis Groningen, Groningen, Netherlands
- Starship Children's Hospital, Auckland, New Zealand
- Puerto Rico (2):
  - University of Puerto Rico School of Medicine Medical Sciences Campus, San Juan
  - San Jorge Childrens Hospital, Santurce
- Switzerland (3):
  - Swiss Pediatric Oncology Group Bern, Bern
  - Swiss Pediatric Oncology Group Geneva, Geneva
  - Swiss Pediatric Oncology Group Lausanne, Lausanne

REFERENCES:
- [Result] Kuttesch JF Jr, Krailo MD, Madden T, Johansen M, Bleyer A; Children's Oncology Group. Phase II evaluation of intravenous vinorelbine (Navelbine) in recurrent or refractory pediatric malignancies: a Children's Oncology Group study. Pediatr Blood Cancer. 2009 Oct;53(4):590-3. doi: 10.1002/pbc.22133. PMID 19533657